CLINICAL TRIAL: NCT05075499
Title: LONGEVITY OF IMMUNE RESPONSE TO COVID-19 VACCINE IN VACCINATED MULTIPLE SCLEROSIS PATIENTS TREATED WITH TERIFLUNOMIDE (AUBAGIO) OR ALEMTUZUMAB (LEMTRADA)
Brief Title: Immune Response to COVID-19 Vaccine in Multiple Sclerosis Patients Treated With Teriflunomide and Alemtuzumab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Prof. Anat Achiron, Director, Multiple Sclerosis Center, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8182-21 SMC
Record Dates: First submitted 2021-10-06; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; COVID-19; Vaccination; Teriflunomide (Aubagio); Alemtuzumab (Lemtrada); Immune responses; IgG; B-cells; T-cells
MeSH Terms: conditions — Multiple Sclerosis; COVID-19 | interventions — heterologous prime boost COVID-19 vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MS no immunomodulatory treatment (Active Comparator): MS patients receiving no immunomodulatory treatment
  Interventions: Biological: COVID-19 vaccination
- MS Teriflunomide treatment (Active Comparator): MS patients under treatment with Teriflunomide
  Interventions: Biological: COVID-19 vaccination
- MS Alemtuzumab treatment (Active Comparator): MS patients under treatment with Alemtuzumab
  Interventions: Biological: COVID-19 vaccination

INTERVENTIONS:
Biological: COVID-19 vaccination — Blood sample obtained before, 1 , 3 and 6 months after the intervention
  Other Names: Blood withdrawn

SUMMARY:
Phase IV, 3-armed, prospective, open-label, single-center, Israeli study, examining the response to SARS-CoV-2 vaccination in 30 teriflunomide-, 10 alemtuzumab-treated patients, and 30 age-matched (for the teriflunomide group) untreated MS patients. Treatments will be administered according to common local practice. Demographic, clinical, treatment-related and COVID-19-related data will be collected. Blood samples will be drawn for each participant at baseline (before COVID-19 vaccination), and at 1, 3, 6, (and possibly 12) months post 2nd dose of COVID-19 vaccine. Humoral, B-cell and T-cell responses will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

(1) Diagnosis of multiple sclerosis (MS) according to 2017 McDonald criteria. (2) Age >=18 years.

(3) Treatment with Teriflunomide for at least 6 months/or 4 to 18 months after the last course treatment with Alemtuzumab/or untreated.

(4) Signed written informed consent.

Exclusion Criteria:

(1) Cognitive decline that precludes understanding the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Percent of SARS-COV-2 antibody positive MS COVID-19 vaccinees at 1-month post 2nd COVID-19 vaccine dose. | 6 months
  Detection of SARS-CoV-2 IgG antibodies in blood samples will be performed using Euroimmun (EI, Lubeck, Germany) anti-SARS-CoV-2 IgG quantitative ELISA kit based on a recombinant S1 subunit of the SARS-CoV-2 spike protein

SECONDARY OUTCOMES:
Percent of SARS-COV-2 antibody positive MS COVID-19 vaccinees at 3 and 6 months post 2nd COVID-19 vaccination. | 12months
  Detection of SARS-CoV-2 IgG antibodies in blood samples will be performed using Euroimmun (EI, Lubeck, Germany) anti-SARS-CoV-2 IgG quantitative ELISA kit based on a recombinant S1 subunit of the SARS-CoV-2 spike protein
SARS-COV-2 antibody titer at 1,3 and 6 months post 2nd COVID-19 vaccination. | 12 months
  Detection of SARS-CoV-2 IgG antibodies in blood samples will be performed using Euroimmun (EI, Lubeck, Germany) anti-SARS-CoV-2 IgG quantitative ELISA kit based on a recombinant S1 subunit of the SARS-CoV-2 spike protein
SARS-COV-2 B-cell memory response at 1,3 and 6 months post 2nd COVID-19 vaccination. | 12 months
  Reversed antigen human IgG SARS-CoV-2 receptor-binding domain (RBD) ELISpotPLUS will be used according to the manufacturer instructions.
Percent of MS COVID-19 vaccinees with SARS-COV-2 T-cell memory positive response at 1,3 and 6 months post 2nd COVID-19 vaccination. | 12 months
  Positive T cell response will be calculated according to the highest number of IFN-γ/IL-2 secreting cells in the FluoroSpot
SARS-COV-2 T-cell memory response at 1,3 and 6 months post 2nd COVID-19 vaccination. | 12 months
  As indicated in outcome #5
Percent of MS COVID-19 vaccinees with positive double immune response (two responses of the possible three), or positive triple immune response (IgG, T-cell and B-cell memory positive) at 6 months post 2nd COVID-19 vaccination. | 6 months
  Statistical analysis
Percent of MS COVID-19 vaccinees with SARS-COV-2 B-cell memory positive response at 1,3 and 6 months post 2nd COVID-19 vaccination. Positive cut-off value will be determined as higher than 10 SFU. | 6 months
  Statistical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol: PMID — http://pubmed.ncbi.nlm.nih.gov/32532623/ — Study scientific background
- Available data/document: Study Protocol: PMID — http://apps.who.int/iris/handle/10665/338671 — Study scientific background. World Health Organization 2021. Background document on mRNA vaccine BNT162b2 (Pfizer-BioNTech) against COVID-19.
- Available data/document: Study Protocol: PMID — http://pubmed.ncbi.nlm.nih.gov/32727835/ — Study scientific background.
- Available data/document: Study Protocol: PMID — http://pubmed.ncbi.nlm.nih.gov/32769063/ — Study scientific background.
- Available data/document: Study Protocol: PMID — http://pubmed.ncbi.nlm.nih.gov/25636714/ — Study scientific background.
- Available data/document: Study Protocol: PMID — http://pubmed.ncbi.nlm.nih.gov/24444048/ — Alemtuzumab medication
- Available data/document: Study Protocol: PMID — https://pubmed.ncbi.nlm.nih.gov/27766281/ — Alemtuzumab medication
- Available data/document: Study Protocol: PMID — https://pubmed.ncbi.nlm.nih.gov/31898276/ — Alemtuzumab medication
- Available data/document: Study Protocol: PMID — http://products.sanofi.us/aubagio/aubagio.html — Aubagio (teriflunomide) [prescribing information]. Cambridge (MA): Genzyme Corporation; September 2012.
- Available data/document: Study Protocol: PMID — http://pubmed.ncbi.nlm.nih.gov/31898276/ — Aubagio (teriflunomide) medication
- Available data/document: Study Protocol: PMID — http://pubmed.ncbi.nlm.nih.gov/29275977/ — Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria.